CLINICAL TRIAL: NCT07375264
Title: Long-term Outcomes of Ultrasound-guided Percutaneous Bilateral Cardiac Sympathetic Denervation in Patients With Refractory Arrhythmic Storm: a Single-center Case Series
Brief Title: Cardiac Sympathetic Denervation in Patients With Refractory Arrhythmic Storm: a Single-center Case Series
Status: Completed | Type: Observational
Sponsor: Jose Manuel López González (Other)
Responsible Party: Sponsor-Investigator, Jose Manuel López González, MD. Consultant Anesthesiologist and Pain Physician, Fundación para la Investigación Biosanitaria del Principado de Asturias
Organization: Fundación para la Investigación Biosanitaria del Principado de Asturias (Other)
Other Study IDs: 2023/139
Record Dates: First submitted 2026-01-21; First posted 2026-01-29 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Ventricular Arrhythmias; Electrical Storm; Stellate Ganglion Block
Keywords: Stellate ganglion block; Cardiac sympathetic denervation; Electrical storm; Ventricular arrhythmias

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SGB + BCSD.: Patients with arrhythmic storm refractory to conservative medical treatment undergoing stellate ganglion block (SGB) and bilateral cardiac sympathetic denervation (BCSD) for arrhythmic storm control.
  Interventions: Procedure: Cardiac sympathetic denervation.

INTERVENTIONS:
Procedure: Cardiac sympathetic denervation. — Patients underwent stellate ganglion block with 10 ml of levobupivacaine 0.25% and subsequently ultrasound-guided percutaneous bilateral cardiac sympathetic denervation , two neuroablative lesions were created using conventional radiofrequency treatment at 60°C, 20 V for 90 seconds.

SUMMARY:
The objective of our study was to evaluate the effectiveness of stellate ganglion block (SGB) and of the bilateral cardiac sympathetic denervation (BCSD) in patients with electrical storm refractory to conventional treatment..

DETAILED DESCRIPTION:
A prospective, single-center observational study was designed with the aim of evaluate the safety and short-term efficacy of SGB within the first 24 hours, as well as the long-term effectiveness of ultrasound-guided percutaneous BCSD at 12 months, in patients with refractory electrical storm.

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 years of age.
* arrhythmic storm refractory to conventional treatment.

Exclusion Criteria:

* patients younger than 18 years of age.
* previous history of heart transplantation.
* history of previous surgical cardiac sympathetic denervation.
* patients with neck anatomy considered unsuitable for the procedure (including previous neck surgery, burns, the presence of extensive scars, or large goiters with significant displacement of adjacent structures).
* contraindications to the interventional technique (such as infection at the puncture site, or refusal to provide consent).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: After approval of the study by Principality of Asturias Drug Research Ethics Committee (CEImPA), Spain and obtaining informed consent from the participants, all consecutive patients who underwent SGB followed by BCSD as part of the treatment for refractory electrical storm were included.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2023-04-11 (Actual); Primary Completion 2025-01-13 (Actual); Study Completion 2025-12-15 (Actual)

PRIMARY OUTCOMES:
Arrhythmic burden. | The arrhythmic burden was assessed both in the early period (first 24 hours following SGB) and in the long term (during the 12 months following BCSD).
  The arrhythmic burden was quantified by the number of sustained ventricular arrhythmias, antitachycardia pacing (ATP) therapies, and ICD (implantable cardioverter-defibrillator) shocks recorded during the follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel García Iglesias, MD.PhD, Principal Investigator — Central University Hospital of Asturias, 33001, Spain
Locations (1):
- FINBA, Oviedo, Principality of Asturias, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Jentzer JC, Noseworthy PA, Kashou AH, May AM, Chrispin J, Kabra R, Arps K, Blumer V, Tisdale JE, Solomon MA; American College of Cardiology Critical Care Cardiology and Electrophysiology Sections. Multidisciplinary Critical Care Management of Electrical Storm: JACC State-of-the-Art Review. J Am Coll Cardiol. 2023 Jun 6;81(22):2189-2206. doi: 10.1016/j.jacc.2023.03.424. PMID 37257955
- [Result] Zeppenfeld K, Tfelt-Hansen J, de Riva M, Winkel BG, Behr ER, Blom NA, Charron P, Corrado D, Dagres N, de Chillou C, Eckardt L, Friede T, Haugaa KH, Hocini M, Lambiase PD, Marijon E, Merino JL, Peichl P, Priori SG, Reichlin T, Schulz-Menger J, Sticherling C, Tzeis S, Verstrael A, Volterrani M; ESC Scientific Document Group. 2022 ESC Guidelines for the management of patients with ventricular arrhythmias and the prevention of sudden cardiac death. Eur Heart J. 2022 Oct 21;43(40):3997-4126. doi: 10.1093/eurheartj/ehac262. No abstract available. PMID 36017572
- [Result] Gao D, Sapp JL. Electrical storm: definitions, clinical importance, and treatment. Curr Opin Cardiol. 2013 Jan;28(1):72-9. doi: 10.1097/HCO.0b013e32835b59db. PMID 23160339
- [Result] Baldi E, Dusi V, Rordorf R, Currao A, Compagnoni S, Sanzo A, Gentile FR, Frea S, Gravinese C, Angelini F, Cauti FM, Iannopollo G, De Sensi F, Gandolfi E, Frigerio L, Crea P, Zagari D, Casula M, Binaghi G, Sangiorgi G, Barone L, Persampieri S, Dell'Era G, Patti G, Colombo C, Mugnai G, Tavella D, Notaristefano F, Barengo A, Falcetti R, Girardengo G, D'Angelo G, Tanese N, Sgromo V, De Ferrari GM, Savastano S; all the STAR study group. Efficacy of early use of percutaneous stellate ganglion block for electrical storms. Eur Heart J Acute Cardiovasc Care. 2024 Dec 3;13(11):757-765. doi: 10.1093/ehjacc/zuae109. PMID 39317656
- [Result] Savastano S, Baldi E, Compagnoni S, Rordorf R, Sanzo A, Gentile FR, Dusi V, Frea S, Gravinese C, Cauti FM, Iannopollo G, De Sensi F, Gandolfi E, Frigerio L, Crea P, Zagari D, Casula M, Sangiorgi G, Persampieri S, Dell'Era G, Patti G, Colombo C, Mugnai G, Notaristefano F, Barengo A, Falcetti R, Perego GB, D'Angelo G, Tanese N, Currao A, Sgromo V, De Ferrari GM; STAR study group. Electrical storm treatment by percutaneous stellate ganglion block: the STAR study. Eur Heart J. 2024 Mar 7;45(10):823-833. doi: 10.1093/eurheartj/ehae021. PMID 38289867
- [Result] Patel RA, Condrey JM, George RM, Wolf BJ, Wilson SH. Stellate ganglion block catheters for refractory electrical storm: a retrospective cohort and care pathway. Reg Anesth Pain Med. 2023 May;48(5):224-228. doi: 10.1136/rapm-2022-104172. Epub 2023 Feb 1. PMID 36725213
- [Result] Baldi E, Conte G, Zeppenfeld K, Lenarczyk R, Guerra JM, Farkowski MM, de Asmundis C, Boveda S. Contemporary management of ventricular electrical storm in Europe: results of a European Heart Rhythm Association Survey. Europace. 2023 Apr 15;25(4):1277-1283. doi: 10.1093/europace/euac151. PMID 36196613

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-04-11): https://cdn.clinicaltrials.gov/large-docs/64/NCT07375264/Prot_SAP_ICF_000.pdf